CLINICAL TRIAL: NCT00105079
Title: A 48-week, Randomized, Open-label, 2-arm Study to Compare the Efficacy of Saquinavir/Ritonavir Twice Daily (BID) Plus Emtricitabine/Tenofovir Once Daily (QD) Versus Lopinavir/Ritonavir BID Plus Emtricitabine/Tenofovir QD in Treatment-naïve Human Immunodeficiency Virus Type 1 (HIV-1) Infected Patients (GEMINI Study)
Brief Title: GEMINI Study - A Study of Saquinavir/Ritonavir in Treatment-Naive Patients With HIV-1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18413
Record Dates: First submitted 2005-03-04; First posted 2005-03-07 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir; Lopinavir; lopinavir-ritonavir drug combination; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Ritonavir

ARMS (2):
- saquinavir/ritonavir (Experimental): saquinavir mesylate 1000 mg twice daily (BID) + ritonavir 100 mg BID + emtricitabine/tenofovir disoproxil fumarate 200/300 mg orally every day for 48 weeks.
  Interventions: Drug: saquinavir [Invirase]; Drug: Emtricitabine/tenofovir disoproxil fumarate; Drug: Ritonavir
- lopinavir/ritonavir (Active Comparator): lopinavir/ritonavir 400/100 mg BID + emtricitabine/tenofovir disoproxil fumarate 200/300 mg orally every day for 48 weeks.
  Interventions: Drug: Lopinavir/ritonavir; Drug: Emtricitabine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: saquinavir [Invirase] — 1000 milligram (mg) Oral (po) twice daily (bid)
  Other Names: Invirase
  Arms: saquinavir/ritonavir
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir 400/100 mg po bid
  Other Names: Kaletra
  Arms: lopinavir/ritonavir
Drug: Emtricitabine/tenofovir disoproxil fumarate — Emtricitabine/tenofovir disoproxil fumarate 200/300 mg po qd
  Other Names: Truvada
Drug: Ritonavir — 100 mg po bid
  Other Names: Norvir
  Arms: saquinavir/ritonavir

SUMMARY:
This 2 arm study will evaluate the efficacy, safety and tolerability of saquinavir/ritonavir or lopinavir/ritonavir in combination with emtricitabine/tenofovir in patients with human immunodeficiency virus type 1 (HIV-1) infection who have received no prior HIV treatment. Patients will be randomized to receive either saquinavir/ritonavir 1000/100mg oral (po) twice daily (bid) + emtricitabine/tenofovir 200/300mg po once daily (qd), or lopinavir/ritonavir 400/100mg po bid + emtricitabine/tenofovir 200/300mg po qd. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic HIV-1 infection;
* treatment-naive;
* HIV-1 RNA viral load >=10,000copies/mL;
* women of childbearing potential must have a negative pregnancy test, and must use reliable contraception for the duration of the study and for 90 days after the last dose of study medication.

Exclusion Criteria:

* females who are pregnant or breastfeeding;
* active hepatitis B infection;
* previous treatment with antiretroviral medication;
* patients who have received an investigational drug within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2005-04; Primary Completion 2007-08 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (19):
  - Hobson City, Alabama
  - Tucson, Arizona
  - Berkeley, California
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Ypsilanti, Michigan
  - St Louis, Missouri
  - Newark, New Jersey
  - New York, New York
  - Huntersville, North Carolina
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Canada (4):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (11):
  - Avignon
  - Lyon
  - Marseille
  - Nantes
  - Nice
  - Paris
  - Rouen
  - Strasbourg
  - Suresnes
  - Toulouse
  - Tourcoing
- Ponce, Puerto Rico
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 28 April 2005 and 24 August 2007 at 38 study centers in the United States, Canada, France and Thailand. Patients were randomized to receive saquinavir/ritonavir 1000/100 mg PO BID plus emtricitabine/tenofovir 200/300 mg PO QD or lopinavir/ritonavir 400/100 mg PO BID plus emtricitabine/tenofovir 200/300 mg PO QD .
Period: Overall Study
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Started | 167 | 170
Safety Population | 163 | 168
Completed | 128 | 135
Not Completed | 39 | 35
Not completed — Adverse Event | 5 | 12
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 12 | 12
Not completed — Lack of Efficacy | 9 | 3
Not completed — Refused treatment | 6 | 4
Not completed — Violation of selection criteria at entry | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir | Total
Number analyzed (Participants) | 167 | 170 | 337
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (9.31) | 37.9 (9.60) | 38.1 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 136 | 131 | 267

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) Viral Load <50 Copies/mL
Description: The primary objective of this study was to evaluate the efficacy of saquinavir/ritonavir BID plus emtricitabine/tenofovir QD versus lopinavir/ritonavir BID plus emtricitabine/tenofovir QD in treatment-naïve HIV-1 infected adults.
  Blood samples for HIV-1 RNA viral load measurement were collected at the Week 48 clinic visit. The number of participants with HIV-1 RNA results <50 copies/mL is reported.
Time Frame: Week 48
Population: intent-to-treat (ITT) Population
Measure: Number; unit: participants
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 167 | 170
participants
  Pts. with HIV-1 RNA Viral Load <50 copies/mL - YES | 108 | 108
  Pts. with HIV-1 RNA Viral Load <50 copies/mL - NO | 59 | 62

2. Secondary Outcome: Number of Patients With HIV-1 RNA Viral Load <50 and <400 Copies/mL
Description: The secondary objectives of the study were to evaluate the safety, adherence, and tolerability of saquinavir/ritonavir BID plus emtricitabine/tenofovir QD versus lopinavir/ritonavir BID plus emtricitabine/tenofovir QD in treatment-naïve HIV-1 infected adults.
  Blood samples for HIV-1 RNA viral load measurement were collected at the Week 48 clinic visit. The number of participants with HIV-1 RNA results <50 copies/mL and the number of participants with HIV-1 RNA results <400 copies/mL are reported.
Time Frame: Week 48
Population: Intent-to-Treat Population
Measure: Number; unit: participants
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 167 | 170
participants
  Patients with <50 Copies/mL | 108 [57.4 to 71.9] | 108 [56.3 to 70.8]
  Patients with <400 Copies/mL | 121 [65.7 to 79.2] | 127 [68.2 to 81.2]

3. Secondary Outcome: Change From Baseline in HIV-1 RNA Viral Load
Description: Descriptive statistics for change from baseline in log10 transformed plasma HIV-1 RNA load (copies/mL) were presented by treatment arm. Logarithmic transformation (base 10) was applied to HIV-1 RNA viral load at baseline and at each study visit. Change from baseline in plasma HIV-1 RNA was derived as follows: Change from baseline = Log10 (HIV-1 RNA at week x) - Log10 (HIV-1 RNA at baseline)
Time Frame: Baseline to Week 48
Population: ITT Population. (n) in each of the categories is the number of participants from the ITT population who had data available at that time point.
Measure: Mean (95% Confidence Interval); unit: copies/mL
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 167 | 170
copies/mL
  Baseline | 5.20 [5.1 to 5.3] | 5.17 [5.1 to 5.3]
  Week 48 (n=126,133) | 1.80 [1.8 to 1.9] | 1.83 [1.8 to 1.9]
  Change from Baseline to Week 48 (n=126,133) | -3.39 [-3.5 to -3.3] | -3.36 [-3.5 to -3.2]

4. Secondary Outcome: Change From Baseline in Cluster Differentiation Antigen 4 Positive (CD4+) Lymphocyte Count
Description: Summary statistics for change from baseline in CD4+ lymphocyte count were presented by treatment arm. Change from baseline in CD4+ lymphocyte count was derived as follows: Change from baseline = (CD4+ count at week x) - (CD4+ count at baseline).
Time Frame: Baseline to Week 48
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 167 | 170
cells/mm^3
  Baseline (n=166,169) | 141.5 [108.0 to 168.0] | 142.0 [116.0 to 187.0]
  Week 48 (n=122,131) | 319.0 [277.0 to 370.0] | 348.0 [317.0 to 401.0]
  Change from Baseline to Week 48 (n=121,130) | 178.0 [159.0 to 213.0] | 204.0 [182.0 to 222.0]

5. Secondary Outcome: Number of Participants Assessed for Adverse Events (AEs)
Description: Detailed information for Adverse Events and Serious Adverse Events will be represented in the SAE/AE section of PRS.
Time Frame: reported up to 28 days after the last dose of study treatment. (Up to 52 weeks)
Population: Safety population included all randomized patients who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 163 | 168
participants | 163 | 168

6. Secondary Outcome: Number of Patients Who Discontinued Treatment Due to Abnormal Laboratory Parameters
Description: Routine clinical testing, including hematology and standard chemistry panel was performed at all study visits. Laboratory tests for a fasting lipid profile and fasting insulin determination were obtained at baseline, weeks 24 and 48, and the 4-week follow-up visit. The number of participants who discontinued treatment due to an abnormal laboratory result at any visit is reported.
Time Frame: baseline and all study visits (Up to Week 52)
Population: Safety population included all randomized patients who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Number analyzed (Participants) | 163 | 168
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All new nonserious AEs and SAEs, irrespective of causal relationship, were reported up to 28 days after the last dose of study treatment. Serious AEs considered related to the test drug were to be reported indefinitely. (Up to 52 weeks)
Description: The safety population included all randomized patients who took at least 1 dose of the trial medication and had at least 1 post-baseline safety assessment.
Arm/Group | Saquinavir/Ritonavir | Lopinavir/Ritonavir
Serious Adverse Events (participants affected / at risk) | 24/163 | 19/168
Other Adverse Events (participants affected / at risk) | 76/163 | 92/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saquinavir/Ritonavir (N=163) | Lopinavir/Ritonavir (N=168)
Cerebral toxoplasmosis (Infections and infestations) | 0 | 2
Bronchitis viral (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Cytomegalovirus oesophagitis (Infections and infestations) | 1 | 0
Encephalitis cytomegalovirus (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Toxoplasmosis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Drowning (General disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Victim of crime (Social circumstances) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saquinavir/Ritonavir (N=163) | Lopinavir/Ritonavir (N=168)
Upper respiratory tract infection (Infections and infestations) | 11 | 23
Bronchitis (Infections and infestations) | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 46 | 77
Nausea (Gastrointestinal disorders) | 40 | 55
Vomiting (Gastrointestinal disorders) | 21 | 28
Fatigue (General disorders) | 15 | 12
Headache (Nervous system disorders) | 8 | 14
DIZZINESS (Nervous system disorders) | 12 | 14
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 | 8
INSOMNIA (Psychiatric disorders) | 6 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.